CLINICAL TRIAL: NCT06546475
Title: Tapering Antipsychotics in Patients With Remitted Psychosis: From Bedside to Bench Employing Animal Model and N-Acetylcysteine Study and Back to Bedside
Brief Title: A Pilot Trial of Tapering Antipsychotics for Patients in Remitted Psychosis Co-administering With N-Acetylcysteine
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202401210MIND; NSTC 113-2314-B-002-184-MY3 (Other Grant/Funding Number: National Science and Technology Council (NSTC), Taiwan)
Record Dates: First submitted 2024-07-29; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Psychosis
Keywords: antipsychotic; N-Acetylcysteine; pilot trial; psychosis; relapse; remission; schizophrenia; tapering
MeSH Terms: conditions — Psychotic Disorders; Recurrence; Schizophrenia | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAC add-on 1 (Experimental): NAC add-on with 1200 mg/d
  Interventions: Drug: N-Acetylcysteine
- NAC add-on 2 (Active Comparator): NAC add-on with 2400 mg/d
  Interventions: Drug: N-Acetylcysteine

INTERVENTIONS:
Drug: N-Acetylcysteine — regular dose or high dose add-on
  Other Names: N-Acetylcysteine 2400 mg/d

SUMMARY:
The investigators are going to observe if add-on of n-acetylcysteine (NAC) 1200 or 2400 mg/d during tapering of antipsychotics in patients with remitted psychosis can help to reduce the pre-requisite of stabilization to 3 months (compared to the 6 months prerequisite of a previous Guided Antipsychotic Reduction to Minimum Effective Dose (GARMED) trial,) smoothly, without increased risk of relapse or frequency of adverse events compared to the 2-year results of the GARMED trial

DETAILED DESCRIPTION:
Trial procedure

* Pretreatment: more instructions were delivered regarding the extent and the tempo of dose reduction, warning signal of relapse, timing to call for help if in need to resume rescue dose, and a shared decision-making process during tapering. Pre-treatment of NAC 1200 mg/d will be given for 1-2 weeks and then titrated up to 2400 mg/d to test tolerability. Patients will stay at either dose throughout the remaining of the course as preferable.
* Dose tapering schedule: In the beginning, no more than one-quarter of the baseline antipsychotic dose will be reduced at a time. Patients need to be monitored every 4 weeks (or 1 month) by phone or in person. If they can maintain stabilized for 12 weeks (or 3 months) in a reduced dose, they can take next tapering of no more than one quarter of their current dose again, yielding 9/16 (3/4x3/4) of baseline dose. The subsequent dose reduction will be a reiteration of the previous step, cutting off one-quarter of the current dose following the formula (3/4) powered by n, rather than cutting off another 1/4 of the initial dose. The processes will be reiterated for 4 steps for one year.
* Conditions during tapering: Noteworthily, when the patient is eligible to consider next dose reduction, he or she is empowered to take shared decision-making as they might opt to stay at their current dose for a more extended time for any reason. Patients can reach the study team during the course whenever they felt unsure if any relapse sign might be re-emerging. As needed use of benzodiazepines or hypnotics will be allowed to help control suspected signs of relapse. Patients will be supervised to stay at current dose for a longer term or even re-escalate to previous higher dose if any sign of suspected relapse re-emerges, and then will be closely monitored if their symptoms can be stabilized within 2 weeks.
* Defining relapse: If a patient's recurrent psychotic symptoms cannot be controlled (any PANSS score > 3 in P1, P2, P3, G5, or G9) within 2 weeks under an antipsychotic dose equal to their baseline dose, the patient will be designated as having a relapse.
* Practicability of dosing: The actual dose taken would not always be precisely the number calculated by the formula (3/4)n, as it was impractical to cut off a quarter or even smaller piece of a tablet for daily dosing. Several versions of intermittent or irregular dosing schedules have been generated to meet the needs.
* Extent of dose reduction: The percentage of doses reduced at a designated time point will be calculated by the following formula: [1- (current dose)/(baseline dose)]x100%.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female outpatients or patients at psychiatric daycare service
2. Age 18-60 years old at the time of screening
3. A diagnosis of schizophrenia, schizophreniform disorder, psychosis NOS, based on the DSM-5 criteria
4. With a Positive and Negative Syndrome Scale (PANSS), score < 3 in all 3 positive symptoms (P1: delusion, P2: conceptual disorganization, P3: hallucination) and 2 general symptoms (G9: unusual thought, G5: mannerism and posturing) for at least 3 months
5. With a PANSS score < 4 in all 3 negative symptoms (N1: blunted affect, N4: social withdrawal, N6: lack of spontaneity/flow in conversation) for at least 3 months
6. Currently receiving antipsychotic treatment at a fixed dose for at least 3 months, including long-acting injectable antipsychotic
7. No revised use of benzodiazepines, antidepressants, anticholinergics, or other concomitant medications during the past 3 months

Exclusion Criteria:

1. A score of 5 or more on any of the 30 PANSS rating items at screening
2. Admission to the acute psychiatric unit during the past 6 months
3. A change in dose of current antipsychotic medication in recent 3 months
4. Concomitant use of mood stabilizers, such as lithium, valproic acid, or other anti-epileptic drugs
5. Mental retardation known as IQ below 70 prior to the diagnosis of schizophrenia
6. A history of pervasive mental disorder or bipolar disorder
7. A medical condition with significant cognitive sequelae
8. A history of substance dependence during the past 6 months
9. Currently in pregnancy or breastfeeding
10. A history of allergy to N-Acetylcysteine
11. Patient with phenylketonuria ( because the Actein Effervescent Tablet 600 mg/tab contains aspartame)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Relapse rate (%) | 1 year
  If a patient's recurrent psychotic symptoms cannot be controlled (any PANSS score > 3 in P1, P2, P3, G5, or G9) within 2 weeks under an antipsychotic dose equal to their baseline dose, the patient will be designated as having a relapse

SECONDARY OUTCOMES:
Extent of dose reduction (%) | 1 year
  The percentage of doses reduced at a designated time point will be calculated by the formula: [1- (current dose)/(baseline dose)]x100%
Clinical severity: symptoms | 1 year
  Positive and Negative Syndrome Scale (PANSS) (1 to 7, 1: normal; 7: profound severity)
Clinical severity: global | 1 year
  Clinical Global Impression of Severity (CGI-S) (1 to 7, 1: no illness; 7: most severe)
Personal and Social Functioning | 1 year
  Personal and Social Performance scale (PSP) (0-100, worst to best)
Self-report of subjective wellbeing | 1 year
  EuroQoL-5D visual analogue scale (EQ-5D-VAS) (0-100, worst to best)
Self-report of Quality of Life | 1 year
  Mandarin Chinese version of the WHOQOL-BREF (1~5, 1: very dissatisfied; 5: very satisfied)

OTHER OUTCOMES:
Qualitative measurements by semi-structured interview | 1 year
  At each time point of shared decision-making regarding whether to taper down dose or not, we will conduct a semi-structure interview to explore patient's key considerations, such as psychosocial issues, soundness of supportive system, and self-assessed risk of relapse, which prompt the patient to feel comfortable about continuing tapering, or to halt at current dose for a longer term.
Self-report of Medication Adherence | 1 year
  5-point Likert scale for medication adherence (1: < 20%; 2: 20~40%; 3: 40~60%; 4: 60~80%; 5: > 80%)
Self-report of Medication Satisfaction | 1 year
  7-point Likert scale for medication satisfaction (1: most dissatisfied; 7: most satisfied)
Adverse events | 1 year
  checklist of Udvalg for Kliniske Undersogelser (UKU) Side-effects Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Chung Liu, MD, PhD, Principal Investigator — National Taiwan University, College of Medicine

IPD SHARING:
Plan to Share IPD: No